CLINICAL TRIAL: NCT05472584
Title: Neural Plasticity by Spinal Cord Stimulation and Training in People With Spinal Cord Injury
Brief Title: Spinal Cord Stimulation and Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ismael Seáñez, Assistant Professor of Biomedical Engineering and Neurosurgery, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202206159
Record Dates: First submitted 2022-07-08; First posted 2022-07-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury, spinal cord stimulation, rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: Non-invasive spinal cord stimulation (Experimental): This arm will receive 30 minutes of transcutaneous spinal cord stimulation as participants rest.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Transcutaneous spinal cord stimulation
- Experimental: Activity-based training (Experimental): This arm will perform 30 minutes of activity-based training using leg movements.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Activity-based training
- Experimental: Activity-based training wtih non-invasive spinal cord stimulation (Experimental): This arm will receive transcutaneous spinal cord stimulation as participants perform 30 minutes of activity-based training using leg movements.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Activity-based training; Other: Transcutaneous spinal cord stimulation
- Experimental: Non-invasive spinal cord stimulation and strength training (Experimental): This arm will receive transcutaneous spinal cord stimulation as participants perform strengthening exercises.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Activity-based training; Other: Transcutaneous spinal cord stimulation
- Experimental: Non-invasive spinal cord stimulation and precision training (Experimental): This arm will receive transcutaneous spinal cord stimulation as participants perform precision-control and dexterity exercises.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Activity-based training; Other: Transcutaneous spinal cord stimulation
- Experimental: Long-term activity-based training with non-invasive spinal cord stimulation (Experimental): This arm will receive 4 weeks of activity-based training with transcutaneous spinal cord stimulation
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Electrophysiology assessment - reticulospinal tract; Other: Electrophysiology assessment - spinal motoneuron; Other: Activity-based training; Other: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Other: Electrophysiology assessment - corticospinal tract — Kinematics and cortical spinal motor excitability
Other: Electrophysiology assessment - reticulospinal tract — Kinematics and reticular spinal motor excitability
Other: Electrophysiology assessment - spinal motoneuron — Kinematics and spinal motoneuron excitability
Other: Activity-based training — Motor task
  Arms: Experimental: Activity-based training; Experimental: Activity-based training wtih non-invasive spinal cord stimulation; Experimental: Long-term activity-based training with non-invasive spinal cord stimulation; Experimental: Non-invasive spinal cord stimulation and precision training; Experimental: Non-invasive spinal cord stimulation and strength training
Other: Transcutaneous spinal cord stimulation — Non-invasive spinal cord stimulation
  Arms: Experimental: Activity-based training wtih non-invasive spinal cord stimulation; Experimental: Long-term activity-based training with non-invasive spinal cord stimulation; Experimental: Non-invasive spinal cord stimulation; Experimental: Non-invasive spinal cord stimulation and precision training; Experimental: Non-invasive spinal cord stimulation and strength training

SUMMARY:
This study will help the investigators better understand the changes in short-term excitability and long-term plasticity of corticospinal, reticulospinal and spinal neural circuits and how the changes impact the improvements of spinal cord stimulation (SCS) mediated motor function.

DETAILED DESCRIPTION:
The goal of this project is to determine the changes in short-term excitability and long-term plasticity of corticospinal, reticulospinal, and spinal neural circuits that are involved in SCS-mediated motor function improvements in individuals with spinal cord injury (SCI). The study will: (1) Determine the short-term effects in neural excitability induced by SCS and activity-based training. (2) Determine the effect of motor training on short-term changes in neural excitability enabled by SCS. (3) Determine the long-term changes in motor control and neural plasticity induced by combined SCS and activity-based training in individuals with chronic SCI. Having a better understanding of the neural mechanisms that are enhanced by SCS can allow the development of therapies that directly target the excitability and plasticity states of these structures towards improved and accelerated recovery.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* Age between 16 and 65 years old
* Healthy people with no major comorbidities of any organ system

Exclusion Criteria:

Healthy Volunteers

* Subjects younger than 16 or older than 65 years old
* Subjects not providing consent or not able to consent
* Subjects with any acute or chronic pain condition
* Subjects with any acute or chronic disease of a major organ system
* Use of analgesics within 24 hours prior to study period
* Use of caffeine with 3 hours of study appointment

Inclusion criteria:

Participants with spinal cord injury (SCI)

* Age between 16-65 years old
* Traumatic SCI C4-T9 level, incomplete (ASIA C or D)
* at least 1 year post injury
* Stable medical condition
* difficulty independently performing leg movements in routine activities
* able to follow simple commands
* able to speak and respond to questions

Exclusion criteria:

Participants with spinal cord injury (SCI)

* Subjects younger than 16 or older than 65 years old
* Not willing or able to provide consent
* Any acute or chronic pain condition
* Any acute or chronic disease of a major organ system
* Use of analgesics within 24 hours prior to study appointment
* Use of caffeine with 3 hours of study appointment
* Presence of tremors, spasms and other significant involuntary movements
* Etiology of SCI other than trauma
* Concomitant neurologic disease traumatic brain injury (TBI) that will significantly impact the ability to follow through on study directions, multiple sclerosis (MS), stroke or peripheral neuropathy)
* History of significant medical illness (cardiovascular disease, uncontrolled diabetes, uncontrolled hypertension, osteoporosis, cancer, chronic obstructive pulmonary disease, severe asthma requiring hospitalization for treatment, renal insufficiency requiring dialysis, autonomic dysreflexia, etc).
* Severe joint contractures disabling or restricting lower limb movements.
* Unhealed fracture, contracture, pressure sore, urinary tract infection or other uncontrolled infections, other illnesses that might interfere with lower extremity exercises or testing activities
* Depression, anxiety, or cognitive impairment
* Deficit of visuospatial orientation
* Sitting tolerance less than 1 hour
* Severe hearing or visual deficiency
* Miss more than 3 appointments without notification
* Unable to comply with any of the procedures in the protocol
* Botulinum toxin injection in lower extremity muscles in the prior six months
* Any passive implants (osteosynthesis material, metallic plates or screws) below T9.
* Any implanted stimulator in the body (pacemaker, vagus nerve stimulator, etc.)
* History of alcoholism or another drug abuse
* Pregnancy (or possible pregnancy)
* Having an Intrathecal Baclofen Therapy Pump (ITB pump)
* History of epilepsy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potentials amplitude and latency | 30 minutes before and 30 minutes after intervention; 4 weeks
  This primary outcome is a measure of changes in corticospinal tract excitability and plasticity as quantified by changes in the amplitude size and onset latency of motor evoked potentials elicited via transcranial magnetic stimulation.
Reaction time to startle response | 30 minutes before and 30 minutes after intervention; 4 weeks
  This primary outcome is a measure of changes in reticulospinal tract excitability after training as quantified by changes in reaction time after a startling auditory stimulus.
F-wave response persistence | 30 minutes before and 30 minutes after intervention; 4 weeks
  This primary outcome is a measure of changes in spinal motoneuron excitability as quantified by changes in the persistence of F-wave responses elicited via peripheral nerve stimulation.

SECONDARY OUTCOMES:
Changes in time to completion from baseline | Baseline, 30 minutes, and 4 weeks
  Participants will perform cursor control as a computer game. This outcome measure is the time it takes participants to complete each task.
Change in movement smoothness | Baseline, 30 minutes, and 4 weeks
  This outcome is a measure of changes in movement smoothness when operating the computer cursor with the body.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Seanez, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States